CLINICAL TRIAL: NCT04190888
Title: Sickle Cell Uric Acid (SCUA) - Cohort Repository
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Other Study IDs: HM20016157
Record Dates: First submitted 2019-12-05; First posted 2019-12-09 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Chronic Kidney Diseases; Sickle Cell Disease
Keywords: Uric acid
MeSH Terms: conditions — Renal Insufficiency, Chronic; Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — Urine and Serum samples will be stored in a research repository
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sickle Cell Disease: Patients with sickle cell disease will be followed prospectively
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention - observational study

SUMMARY:
The purpose of this research is to study the causes of Sickle Cell kidney disease, as well as to collect and store samples and information about people with Sickle Cell Disease.

DETAILED DESCRIPTION:
Sickle Cell Disease causes kidney injury over time, but it is not clear why some individuals have very significant chronic kidney disease and why some do not. The purpose of this research is to study whether having high levels of 'uric acid,' which is a naturally occurring molecule in the body that may increase kidney injury and systemic inflammation, accelerates the progression of chronic kidney disease over time. Researchers will measure the number of participants that have high uric acid levels at the beginning of the study, as well as the number of participants that develop new high levels throughout the study. The study will also try to determine what causes the high uric acid levels in some patients but not others. The results of this study could help understand kidney injury and uric acid in sickle cell disease better.

ELIGIBILITY:
Inclusion Criteria:

* Age 5-29 years
* Sickle cell disease as diagnosed by hemoglobin electrophoresis, or by newborn screen per standard of care
* Currently receiving comprehensive sickle cell care at the Children's Hospital of Richmond at VCU or in the adult Internal Medicine sickle cell care clinic at VCU.

Exclusion Criteria:

* Those who have received organ, stem cell, or bone marrow transplantation. - Those who require chronic dialysis

Ages: 5 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants currently receiving medical care from the pediatric or adult hematology comprehensive sickle cell centers.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Percentage of participants in the sample with hyperuricemia | Baseline
  (i.e. high uric acid levels) out of all patients with a uric acid level measured at baseline.
Incidence rate of hyperuricemia per year | Baseline to year 5
  Calculate the incidence rate of new cases of hyperuricemia per year in each year of the cohort study
The mean rate of change of estimated glomerular filtration rate (eGFR) per year in those with hyperuricemia and those with normouricemia | Baseline to year 5
  Determine the mean rate of change of eGFR per year for each group.

CONTACTS AND LOCATIONS:
Overall Officials: Cristin Kaspar, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes